CLINICAL TRIAL: NCT03483376
Title: Effectiveness of Antimicrobial Photodynamic Therapy for the Elimination of Dental Black Stain: A Randomised Clinical Trial
Brief Title: aPDT for the Remediation of Dental Black Stain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Chirag Sheth, Associate Professor in Epidemiology and Public Health, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VVESES
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Dental Plaque; Tooth Discoloration
Keywords: black stain; dental plaque; antimicrobial photodynamic therapy; curcumin; tooth discoloration
MeSH Terms: conditions — Dental Plaque; Tooth Discoloration | interventions — Dental Prophylaxis

STUDY DESIGN:
Intervention Model Description: Two parallel arms of the study will be used. One arm will receive dental plaque removal using standard protocol. The other arm will receive the standard plaque removal, followed by antimicrobial photodynamic therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dental prophylaxis (Active Comparator): Study volunteers with black plaque stained teeth will receive standard dental prophylactic cleaning to remove the stain. The prophylaxis will be carried out using an ultrasonic scaler, prophylaxis brush and abrasive paste.
  Interventions: Procedure: Dental prophylaxis
- Dental prophylaxis + aPDT (Experimental): Study volunteers with black plaque stained teeth will receive standard dental prophylactic cleaning, followed by antimicrobial photodynamic therapy (aPDT) to remove the stain. The prophylaxis will be carried out using an ultrasonic scaler, prophylaxis brush and abrasive paste. The aPDT protocol is as follows:
  * Patient will rinse the oral cavity with 20 ml of an aqueous solution of curcumin (photosensitizer; 1.5 g/L) for 30 seconds.
  * Blue light from a Bluephase 20i curing lamp will be applied perpendicularly for 1 min per tooth (30 seconds on the vestibular side and 30 seconds on the palatal side).
  * Remaining photosensitizer will be removed using the prophylaxis brush. The aPDT protocol is repeated following a rest period of 10 days.
  Interventions: Procedure: Dental prophylaxis; Device: Antimicrobial photodynamic therapy (aPDT)

INTERVENTIONS:
Procedure: Dental prophylaxis — Determining the effectiveness of dental prophylaxis alone in eliminating dental black stain.
Device: Antimicrobial photodynamic therapy (aPDT) — Establishing the effectiveness of dental prophylaxis combined with antimicrobial photodynamic therapy using blue light and curcumin as the photosensitizing agent in eliminating dental black stain.
  Other Names: Dental prophylaxis + aPDT
  Arms: Dental prophylaxis + aPDT

SUMMARY:
In today's society cosmetic dentistry plays an important role in social relationships and in important aspects of life such as job applications and recruitment processes.

Currently, the only available treatment option for patients suffering from black dental pigmentation of bacterial origin is repetitive professional dental cleanings every two or three months, which involve a significant financial outlay, and have been found to be psychologically detrimental due to the lack of a perceived cure.

These pigmentations are of unknown etiology, although there has been reported the presence of black-pigment producing bacteria, such as Porphyromonas gingivalis, Tannerella forsythia and Aggregatibacter actinomycetemcomitans in such black plaque. These bacteria are found in a group known as periodontopathogens, bacteria responsible for the appearance of periodontitis, an oral chronic disease with high prevalence.

In this context, photodynamic therapy, which uses the application of diode light with a wavelength between 400-500 nm for the elimination of periodontal pathogenic bacteria, has demonstrated effectiveness and absence of adverse effects on the management of patients with periodontitis.

The proposed study seeks to evaluate the effect of photodynamic therapy on teeth with extrinsic black pigment, in order achieve an eradication of the stains. The investigators will also proceed to analyze in depth the bacterial composition of these stains before the application of photodynamic therapy, in order to stablish the aetiological agents of this black plaque.

DETAILED DESCRIPTION:
One of the most common problems facing the dentist in daily practice is the treatment of the chromatic alterations of the teeth, both of extrinsic origin and of intrinsic origin. The former, caused by the incorporation of chromogenic materials into enamel and dentin, either before or after the tooth eruption, require more complex and usually more aggressive treatments in order to eliminate them. On the other hand, the latter, caused by the deposition of pigments or detritus on the tooth surface, are usually removed more easily, causing little or no damage to the enamel.

However, among the latter, black extrinsic dental stains caused by pigmented bacteria represent a clear exception to the rule. These deposits, which manifest in the form of points or lines of black color located parallel to the gingival margin of the teeth in the cervical third, are firmly attached to the enamel, making them very difficult to remove.

Although the exact etiology of the formation of dental black stain due to pigmented bacteria is not clear, it has been suggested that it arises due to the production of a pigment with characteristics similar to protohemin and protoporphyrin by black-pigmented bacteria. The application of light to inactivate and disinfect intraoral sites is gaining interest in the field of dentistry. Antimicrobial photodynamic therapy is defined as the inactivation of cells, microorganisms or molecules induced by light. The mechanism of action of photodynamic therapy is defined as the process by which a photosensitizer (photoactivable substance) is captured by microorganisms and, after exposure to light at an appropriate wavelength, remains in an excited state. The photosensitizer then transfers energy from light to oxygen molecules to generate singlet oxygen and free radicals that are cytotoxic to the cells.

Published studies suggest that antimicrobial photodynamic therapy can effectively reduce the population of microbial pathogens, also presenting the following advantages: absence of phototoxic effect for human cells, possible clinical, microbiological and immunological benefits, rapid and painless application of light, penetration of light into tissues and plaque and, thereby, elimination of bacteria present in gingival epithelial cells, and finally, selectivity towards pathogenic microorganisms.

The main objective of this research is the application of antimicrobial photodynamic therapy in the control of dental black stain caused by pigmented bacteria.

ELIGIBILITY:
Inclusion Criteria:

* volunteers with dental black stain in at least two teeth (non-filled, with partner in the opposite arch)
* volunteers older than 12 years

Exclusion Criteria:

* volunteers receiving antibiotic treatment within the month prior to enrolment

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Area and depth of color of black stain - 6 Months | 6 months post final treatment step for each study arm
  Area and depth of color of black stain 6 months post aPDT - Digital intraoral photographs will be analyzed using image analysis software.

SECONDARY OUTCOMES:
Sensitivity and pain | 24 hours post final treatment step for each study arm
  Dental sensitivity and/or pain following the final treatment step for each study arm, measured by Wong-Baker faces scale. This is a graphic-numeric scale used to allow the patient to describe the sensitivity or pain they are experiencing. It consists of a row of 6 faces arrayed from left to right displaying a range of expressions denoting increased pain. This is accompanied by a numerical scale 0, 2, 4, 6, 8, 10 where 0 is no pain (smiley face) to 10 being the worst pain imaginable (crying, extremely sad face). Below the numerical description, patients may read the descriptions of pain related to each face, ranging from 0 (No Hurt) to 10 (Hurts Worst). Higher scores (right hand side of the scale; sad crying face) indicate higher discomfort or pain, whilst lower scores (left hand side of the scale, happier face) indicate less discomfort or pain. The scale may be applied rapidly and easily facilitating the follow up of patients in a simple, reproducible manner.

OTHER OUTCOMES:
Area and depth of color of black stain - 3 Months | 3 months post final treatment step for each study arm
  Area and depth of color of black stain 3 months post aPDT - Digital intraoral photographs will be analyzed using image analysis software.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Veses, Principal Investigator — Cardenal Herrera University
Locations (1):
- Clinica Odontologica Universitaria CEU, Alfara del Patriarca, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soukos NS, Som S, Abernethy AD, Ruggiero K, Dunham J, Lee C, Doukas AG, Goodson JM. Phototargeting oral black-pigmented bacteria. Antimicrob Agents Chemother. 2005 Apr;49(4):1391-6. doi: 10.1128/AAC.49.4.1391-1396.2005. PMID 15793117
- [Background] Araujo NC, Fontana CR, Gerbi ME, Bagnato VS. Overall-mouth disinfection by photodynamic therapy using curcumin. Photomed Laser Surg. 2012 Feb;30(2):96-101. doi: 10.1089/pho.2011.3053. Epub 2012 Jan 6. PMID 22224655
- [Background] Leite DP, Paolillo FR, Parmesano TN, Fontana CR, Bagnato VS. Effects of photodynamic therapy with blue light and curcumin as mouth rinse for oral disinfection: a randomized controlled trial. Photomed Laser Surg. 2014 Nov;32(11):627-32. doi: 10.1089/pho.2014.3805. Epub 2014 Oct 24. PMID 25343373
- [Background] Carrera ET, Dias HB, Corbi SCT, Marcantonio RAC, Bernardi ACA, Bagnato VS, Hamblin MR, Rastelli ANS. The application of antimicrobial photodynamic therapy (aPDT) in dentistry: a critical review. Laser Phys. 2016 Dec;26(12):123001. doi: 10.1088/1054-660X/26/12/123001. Epub 2016 Nov 9. PMID 29151775